CLINICAL TRIAL: NCT06692673
Title: Use of Linaclotide as a Single Agent Colonoscopy Bowel Preparation Regimen; A Pilot Trial
Brief Title: Linaclotide for Colonoscopy Bowel Prep
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB202400687
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Patients Scheduled for Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients scheduled for Colonoscopy (Experimental): Adult in-patients, 18 years of age and older, scheduled for an in-patient screening or diagnostic colonoscopy
  Interventions: Drug: Use of Linaclotide as a single agent Colonoscopy prep

INTERVENTIONS:
Drug: Use of Linaclotide as a single agent Colonoscopy prep — We plan to conduct a pilot study to determine the feasibility of a quality bowel preparation with two 290mg doses of Linaclotide (first dose given 36 hours before, and the other 8 hours prior to the procedure) along with 2 Liters of Gatorade (to prevent dehydration) given the day prior to the colonoscopy instead of the current standard 4 liters of PEG regimen. All study participants will be asked to consume a clear liquid diet for 24hours before the procedure.
  Other Names: Linaclotide prep

SUMMARY:
The goal of this clinical trial is to learn if drug Linaclotide can be used as a single agent regimen to adequately prepare bowel for colonoscopy.

The main question it aims to answer is:

Does drug Linaclotide with Gatorade provide adequate bowel preparation for colonoscopy instead of the standard 4 Liters of Polyethylene glycol (PEG)?

Participants will:

Take one 290mg dose of Linaclotide 36 hours before the procedure and One 290mg dose of Linaclotide 8 hours before the procedure + 2 Liters of Gatorade and a clear liquid diet 24 hours before the procedure. As per standard of care, all patients will be made Nil Per Oral (NPO) starting midnight before the procedure.

The colonoscopy report will then be reviewed for Boston Bowel Preparation Score (BBPS) as a marker of bowel preparation quality, insertion time as a marker of procedure difficulty as well as noted pathology and any complications or physician noted comments.

DETAILED DESCRIPTION:
Linaclotide is a novel, FDA approved, intestinal prosecretory agent used to treat chronic constipation and irritable bowel syndrome. Linaclotide reduces colonic transit time and increases luminal fluid secretion. Use of Linaclotide in colonoscopy bowel preparation decreased the volume of oral prep required. We hypothesize that Linaclotide can be used as a single agent regimen to adequately prepare bowel for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients (age 18 years to 65) admitted, who are scheduled for a colonoscopy during their admission.

Exclusion Criteria:

* Pregnant patients
* Patients with weight less than 116 pounds
* Patients with prior colon resection surgeries
* Presence of colostomy
* Patients undergoing sigmoidoscopy or pouchoscopy
* Patients unable to swallow pills/tablets
* Patients who would use a G or J feeding tubes to administer medications/preparation regimen
* Patients who are unable to consent for themselves
* Patients with a history of renal failure
* Patients already taking Linaclotide
* Patients who experienced hypersensitivity reactions to Linaclotide in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
BBPS a cutoff 6 or greater | Within 48 hours post Colonoscopy
  Number of participants with Boston Bowel Preparation Scale (BBPS) of 6 or greater

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nordenstam, MD PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States